CLINICAL TRIAL: NCT00241696
Title: Air Pollution, Inflammation, and New Onset Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1308; R01HL076647 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2012-04

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To examine air pollution, inflammation and new onset asthma in a large cohort of children in southern California.

DETAILED DESCRIPTION:
BACKGROUND:

Ambient air pollution is well accepted as a cause of asthma exacerbations, but its role in the etiology of new onset asthma is less clear. Evidence for an etiologic role of ambient air pollutants is emerging from epidemiologic studies; however, the ecologic patterns of increasing asthma prevalence concurrent with decreasing levels of some pollutants have raised questions about the validity of these associations. A better understanding of the biological processes that mediate the effects of ambient air pollution on asthma occurrence is likely to contribute to answering these questions. Chronic oxidative/nitrosative stress and airway inflammation are probably critical processes in asthma etiology and these inter-related processes may mediate the increased asthma risk from air pollution.

This study builds on the existing Asthma Incidence Risk (AIR) study which is an ongoing cohort study consisting of 6000 children with new onset asthma. The children live in 12 communities in Southern California. The communities were chosen to give a range of the key ambient air pollutants of ozone, small particulates, NOx, acid vapors and tailpipe emissions.

DESIGN NARRATIVE:

The study will use exhaled nitric oxide (eNO) to investigate the role of inflammation and oxidative/nitrosative stress in the pathobiology of new onset asthma, with a focus on ambient air pollution and genetic susceptibility. The investigators choose ambient pollutants based on potential contribution to oxidative/nitrosative stress (O3; particulates (PM10 and PM2.5 and their chemical constituents, particle counts, NOx (NO and NO2), acid vapors; and fresh tailpipe emissions). The primary hypotheses to be assessed in the program of research are: 1) children with high ambient air pollution exposures have chronic airway inflammation as indicated by elevated eNO. 2) susceptibility to airway inflammation and oxidative/nitrosative stress from ambient air pollution varies by NOS1, NOS2. NOS3. GSTM1. GSTP1. NQO1, and HO-1 haplotypes and functional variants, and 3) children with chronic airway inflammation as indicated by elevated eNO are at increased risk for new onset asthma. To test these hypotheses, the study builds on the population resource of the Asthma Incidence Risk (AIR) study, an ongoing prospective cohort study of the determinants of new onset asthma in 6000 children in 13 southern California communities, and an extensive program of ambient air pollution exposure characterization in these communities. The investigators will measure eNO using off-line techniques and genotype 3000 children from the AIR cohort. A number of resources will enhance the study, including the Children's Environmental Health Center, the Molecular Biology Core of Southern California Environmental Health Sciences Center, and expertise from the Southern California Particle Center and Supersite.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-08; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gilliland — University of Southern California